CLINICAL TRIAL: NCT01256398
Title: A Phase II Study of Dasatinib (Sprycel®) (NSC #732517) as Primary Therapy Followed by Transplantation for Adults >/= 18 Years With Newly Diagnosed Ph+ Acute Lymphoblastic Leukemia by CALGB, ECOG and SWOG
Brief Title: Dasatinib Followed by Stem Cell Transplant in Treating Older Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02621; NCI-2011-02621 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CALGB 10701/CTSU C10701; CDR0000690286; CALGB-10701 (Other: Alliance for Clinical Trials in Oncology); CALGB-10701 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Acute Lymphoblastic Leukemia; Adult B Acute Lymphoblastic Leukemia With t(9;22)(q34.1;q11.2); BCR-ABL1
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Alemtuzumab; Stem Cell Transplantation; Cyclophosphamide; Cytarabine; Dasatinib; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; etoposide phosphate; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine phosphate; Leucovorin; Melphalan; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegfilgrastim; Tacrolimus; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, transplant) (Experimental): See Detailed Description
  Interventions: Biological: Alemtuzumab; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dasatinib; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Etoposide Phosphate; Biological: Filgrastim; Drug: Fludarabine Phosphate; Procedure: In Vitro-Treated Peripheral Blood Stem Cell Transplantation; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Melphalan; Drug: Mercaptopurine; Drug: Methotrexate; Biological: Pegfilgrastim; Other: Pharmacological Study; Drug: Tacrolimus; Drug: Vincristine Sulfate

INTERVENTIONS:
Biological: Alemtuzumab — Given IV
  Other Names: Anti-CD52 Monoclonal Antibody; Campath; Campath-1H; LDP-03; Lemtrada; MabCampath; Monoclonal Antibody Campath-1H
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo peripheral blood allogeneic HCT
  Other Names: Allogeneic; Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo peripheral blood autologous HCT
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Etoposide Phosphate — Given IV
  Other Names: Etopophos
Biological: Filgrastim — Given SC
  Other Names: Filgrastim-aafi; G-CSF; Neupogen; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Procedure: In Vitro-Treated Peripheral Blood Stem Cell Transplantation — Undergo peripheral blood autologous or allogeneic HCT
  Other Names: in vitro-treated PBPC transplantation; in vitro-treated peripheral blood progenitor cell transplantation
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV or PO
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IT, IV, or PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Biological: Pegfilgrastim — Given SC
  Other Names: Filgrastim SD-01; filgrastim-SD/01; Fulphila; HSP-130; Jinyouli; Neulasta; Neulastim; Nyvepria; PEG-filgrastim; Pegcyte; Pegfilgrastim Biosimilar HSP-130; Pegfilgrastim Biosimilar Nyvepria; Pegfilgrastim Biosimilar Pegcyte; Pegfilgrastim Biosimilar PF-06881894; Pegfilgrastim Biosimilar Udenyca; Pegfilgrastim Biosimilar Ziextenzo; pegfilgrastim-apgf; pegfilgrastim-bmez; pegfilgrastim-cbqv; Pegfilgrastim-jmdb; PF-06881894; SD-01; SD-01 sustained duration G-CSF; Udenyca; Ziextenzo
Other: Pharmacological Study — Correlative studies
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This phase II clinical trial studies how well dasatinib followed by stem cell transplant works in treating older patients with newly diagnosed acute lymphoblastic leukemia. Dasatinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving chemotherapy before a stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. Monoclonal antibodies, such as alemtuzumab, may interfere with the ability of cancer cells to grow and spread. Giving more than one drug (combination chemotherapy) and giving dasatinib together with chemotherapy may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the disease-free survival (DFS) and overall survival (OS) profiles in newly diagnosed patients 18 years or older who have Philadelphia chromosome positive (Ph+) (BCR/(v-abl Abelson murine leukemia viral oncogene homolog [ABL]+) acute lymphoblastic leukemia (ALL) receiving sequential dasatinib followed by allogeneic or autologous hematopoietic cell transplant (HCT) or chemotherapy followed by dasatinib maintenance.

SECONDARY OBJECTIVES:

I. Compare the OS and DFS profiles for each of the three cohorts to those from similar populations from other studies.

II. Determine the ability of dasatinib to produce or maintain a BCR/ABL-negative status, as judged by quantitative-polymerase chain reaction (Q-PCR) following sequential dasatinib, chemotherapy, and HCT.

III. Determine the feasibility of collecting adequate peripheral blood stem cells for autologous HCT following dasatinib therapy and assess for residual Ph+ (BCR/ABL+) cells by Q-PCR.

IV. Study the safety and efficacy of autologous HCT following therapy with dasatinib.

V. Study the safety and efficacy of reduced-intensity preparatory regimen followed by an allogeneic HCT following induction therapy with dasatinib.

VI. Study the safety and efficacy of dasatinib maintenance administered after allogeneic or autologous HCT or chemotherapy.

VII. Correlate plasma and cerebrospinal fluid (CSF) levels of dasatinib when given orally during induction.

OUTLINE: As of 8/21/2014, no new patients may be enrolled on E3903.

REMISSION INDUCTION THERAPY (RIT): Patients receive dasatinib orally (PO) daily continuously and dexamethasone PO or intravenously (IV) on days 1-7.

EARLY INTENSIFICATION THERAPY: Patients with bone marrow =< 20% blasts are assigned to cohort A and patients with bone marrow > 20% blasts are assigned to cohort B.

COHORT A: Patients receive dasatinib and dexamethasone as in RIT.

COHORT B: Patients receive dasatinib and dexamethasone as in RIT, and vincristine sulfate IV and daunorubicin hydrochloride IV on days 1, 8, and 15. Patients who do NOT achieve a complete response (CR) or CR with incomplete hematologic recovery based on bone marrow continue on to second induction therapy; patients who achieve a hematologic and morphologic CR continue on to CNS prophylaxis therapy.

SECOND INDUCTION THERAPY: Patients receive dasatinib and dexamethasone as in RIT, cyclophosphamide IV on day 1, daunorubicin hydrochloride IV and vincristine sulfate IV on days 1 and 8, and filgrastim subcutaneously (SC) beginning on day 9 and continuing for >= 7 days or one dose of pegfilgrastim on day 9.

CNS PROPHYLAXIS THERAPY: Patients receive dasatinib PO daily continuously during CNS prophylaxis therapy; methotrexate intrathecally (IT), vincristine sulfate IV, and methotrexate IV over 3 hours on days 1, 15, and 29; methotrexate PO every 6 hours for a total of 4 doses each on days 1-2, 15-16, and 29-30; leucovorin calcium IV on days 2, 16, and 30; and leucovorin PO calcium every 6 hours for a total of 8 doses each on days 3-4, 17-18, and 31-32.

TRANSPLANTATION OR ALTERNATIVE CHEMOTHERAPY AND MAINTENANCE THERAPY: Patients aged 50-70 years with an HLA-matched related or unrelated donor are assigned to allogeneic transplantation, patients aged 50-70 years without an HLA-matched related or unrelated donor are assigned to autologous transplantation, and patients aged > 70 years or who are not transplantation candidates are assigned to alternative chemotherapy.

ALLOGENEIC TRANSPLANTATION: Patients receive fludarabine phosphate IV over 30 minutes and alemtuzumab IV over 30 minutes on days -7 through -3 and melphalan IV over 30 minutes on day -2. Patients undergo allogeneic peripheral blood stem cell transplantation (PBSCT) on day 0. Patients then receive filgrastim SC beginning on day 1 and continuing until count recovery and tacrolimus IV or PO beginning on day -2 and beginning to taper on day 100 (for matched related donors) or day 180 (for mismatched related or unrelated donors). Beginning on day 30, patients receive dasatinib PO daily as maintenance therapy. Treatment continues for >= 12 months in the absence of disease progression.

AUTOLOGOUS TRANSPLANTATION:

MOBILIZATION: Patients receive etoposide phosphate IV continuously on days 1-4, high-dose cytarabine IV over 2 hours every 12 hours for a total of 8 doses on days 1-4, and filgrastim SC once or twice daily beginning on day 14 and continuing until peripheral blood stem cell collection is complete or WBC > 50,000/μL.

LEUKAPHERESIS: Patients undergo leukapheresis beginning when WBC > 10,000/μL for a target collection of >= 5 x 10^6 CD34+ cells/kg. After completion of stem cell collection, patients receive dasatinib PO twice daily until 3 days before transplantation.

TRANSPLANTATION: Beginning >= 4 weeks after recovery from toxicity related to previous treatment, patients receive melphalan IV over 30 minutes on days -2 and -1. Patients undergo autologous PBSCT on day 0. Patients then receive filgrastim SC beginning on day 0 and continuing until count recovery.

MAINTENANCE THERAPY: Beginning on day 30, patients receive dasatinib PO once daily. Treatment continues for >= 12 months in the absence of disease progression.

ALTERNATIVE CHEMOTHERAPY: Beginning 3-10 days after completion of CNS prophylaxis therapy, patients receive etoposide phosphate IV continuously on days 1-4, high-dose cytarabine IV over 2 hours every 12 hours for a total of 8 doses on days 1-4, and filgrastim SC once or twice daily beginning on day 14 and continuing until count recovery.

MAINTENANCE THERAPY: Patients receive dasatinib PO once daily beginning on day 30. Patients also receive vincristine sulfate IV every 4 weeks, dexamethasone for 5 days every 4 weeks, mercaptopurine PO once daily, and methotrexate PO once weekly. Treatment continues for >= 12 months in the absence of disease progression.

NOTE: Patients with CNS leukemia or testicular disease may receive additional treatment.

After completion of study treatment, patients are followed up every month for 1 year, every 3 months for 2 years, every 6 months for 2 years, and every year for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal histologic diagnosis of ALL
* Detection of the t(9;22)(q34;q11) or 3-way variant by metaphase cytogenetics or BCR-ABL positive status by molecular analysis (Q-PCR or fluorescent in situ hybridization [FISH]) in a Cruise Lines International Association (CLIA)-approved laboratory
* No prior therapy except up to one week of corticosteroids and/or hydroxyurea to enable time for the detection of t(9;22)(q34;q11) or BCR/ABL
* Non-pregnant and non-nursing; treatment under this protocol would expose an unborn child to significant risks; women and men of reproductive potential should agree to use an effective means of birth control and contraception should continue for three months after the last dose of dasatinib to allow complete clearance of drug and its principal metabolites from the body; in women of childbearing potential, a pregnancy test will be required at study entry
* Left ventricular ejection fraction >= lower limit of institutional normal
* No myocardial infarction within 6 months
* No ventricular tachyarrhythmia within 6 months
* No major conduction abnormality (unless a cardiac pacemaker is present)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-12-14 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Wieduwilt, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (101):
- United States (101):
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - AdventHealth Orlando, Orlando, Florida
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - The Jewish Hospital, Cincinnati, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming

REFERENCES:
- [Derived] Wieduwilt MJ, Yin J, Wetzler M, Uy GL, Powell BL, Kolitz JE, Liedtke M, Stock W, Beumer JH, Mattison RJ, Storrick E, Christner SM, Lewis LD, Devine S, Stone RM, Larson RA. Dasatinib and dexamethasone followed by hematopoietic cell transplantation for adults with Ph-positive ALL. Blood Adv. 2021 Nov 23;5(22):4691-4700. doi: 10.1182/bloodadvances.2021004813. PMID 34492682

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Chemotherapy, Transplant): All enrolled patients.>
  > Alemtuzumab: Given IV> Allogeneic Hematopoietic Stem Cell Transplantation: Undergo peripheral blood allogeneic HCT> Autologous Hematopoietic Stem Cell Transplantation: Undergo peripheral blood autologous HCT> Cyclophosphamide: Given IV> Cytarabine: Given IV> Dasatinib: Given PO> Daunorubicin Hydrochloride: Given IV> Dexamethasone: Given PO or IV> Etoposide Phosphate: Given IV> Filgrastim: Given SC> Fludarabine Phosphate: Given IV> In Vitro-Treated Peripheral Blood Stem Cell Transplantation: Undergo peripheral blood autologous or allogeneic HCT> Laboratory Biomarker Analysis: Correlative studies> Leucovorin Calcium: Given IV or PO> Melphalan: Given IV> Mercaptopurine: Given PO> Methotrexate: Given IT, IV, or PO> Pegfilgrastim: Given SC> Pharmacological Study: Correlative studies> Tacrolimus: Given IV or PO> Vincristine Sulfate: Given IV
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Transplant)
Started | 66
Completed | 65
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All patients that began treatment.
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 65
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 60.1 [51.2 to 67.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 5

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival Defined From the Date of First Induction Complete Response (CR) to Relapse or Death Due to Any Cause
Description: Estimated using the Kaplan-Meier estimator. Proportions will be estimated using point as well as interval estimators. All interval estimators will be constructed using the finite sample size sampling distribution at the unadjusted two-sided level of 0.05.
Time Frame: At 3 years after CR
Population: All patients that reached CR and chose to continue with the study.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Treatment (Chemotherapy, Transplant): All enrolled patients that reached CR during induction and continued to course 5.>
  > Alemtuzumab: Given IV> Allogeneic Hematopoietic Stem Cell Transplantation: Undergo peripheral blood allogeneic HCT> Autologous Hematopoietic Stem Cell Transplantation: Undergo peripheral blood autologous HCT> Cyclophosphamide: Given IV> Cytarabine: Given IV> Dasatinib: Given PO> Daunorubicin Hydrochloride: Given IV> Dexamethasone: Given PO or IV> Etoposide Phosphate: Given IV> Filgrastim: Given SC> Fludarabine Phosphate: Given IV> In Vitro-Treated Peripheral Blood Stem Cell Transplantation: Undergo peripheral blood autologous or allogeneic HCT> Laboratory Biomarker Analysis: Correlative studies> Leucovorin Calcium: Given IV or PO> Melphalan: Given IV> Mercaptopurine: Given PO> Methotrexate: Given IT, IV, or PO> Pegfilgrastim: Given SC> Pharmacological Study: Correlative studies> Tacrolimus: Given IV or PO> Vincristine Sulfate: Given IV
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 38
percentage of patients | 52.6 [36.8 to 68.5]

2. Secondary Outcome: Probability of Being BCR-ABL Negative in the Bone Marrow and Peripheral Blood at the Completion of the CNS Prophylaxis Course (Restricted to Those Patients Achieving a CR)
Description: Proportions will be estimated based on the combined and individual cohorts.
Time Frame: 10 years
Measure: Number; unit: proportion of participants
Groups:
- Treatment (Chemotherapy, Transplant): All CR patients.
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 64
proportion of participants | 0.667

3. Secondary Outcome: Feasibility of Maintenance Therapy in This Patient Population (Restricted to Those Patients Achieving a CR). Feasibility Will be Defined as the Number of Deaths Ocuring.
Description: Proportions will be estimated based on the combined and individual cohorts.
Time Frame: 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 64
Participants | 5

4. Secondary Outcome: Overall Survival (OS)
Description: as for outcome 1
Time Frame: 10 years
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Treatment (Chemotherapy, Transplant): All enrolled patients.
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 65
Months | 55.9 [31.8 to NA] — Not enough events for upper limit calculation

5. Secondary Outcome: Disease Free Survival (DFS)
Description: as for outcome 1
Time Frame: 10 years
Population: All CR patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 64
Months | 29.7 [21.5 to 43.0]

6. Secondary Outcome: Response
Description: Proportion of patients reaching a CR. A CR requires the following: an absolute neutrophil count (segs and bands) >1000/μL, no circulating blasts, platelets >100,000/μL; adequate bone marrow cellularity with trilineage hematopoiesis, and <5% marrow leukemia blast cells. All previous extramedullary manifestations of disease must be absent (e.g., lymphadenopathy, splenomegaly, skin or gum infiltration, testicular masses, or CNS involvement).
Time Frame: 10 years
Measure: Number; unit: proportion of participants
Arm/Group | Treatment (Chemotherapy, Transplant)
Number analyzed (Participants) | 65
proportion of participants | .9846

ADVERSE EVENTS:
Time Frame: 10 years
Description: This study will utilize the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 to determine the severity of the reaction for adverse event reporting.
Arm/Group | Treatment (Chemotherapy, Transplant)
All-Cause Mortality (participants affected / at risk) | 5/65
Serious Adverse Events (participants affected / at risk) | 5/65
Other Adverse Events (participants affected / at risk) | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Transplant) (N=65)
Multi-organ failure (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Transplant) (N=65)
Anemia (Blood and lymphatic system disorders) | 59 (535)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 4 (5)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 10 (18)
Febrile neutropenia (Blood and lymphatic system disorders) | 27 (41)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 6 (6)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Cardiac disorders - Other, specify (Cardiac disorders) | 6 (9)
Chest pain - cardiac (Cardiac disorders) | 5 (5)
Heart failure (Cardiac disorders) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (4)
Palpitations (Cardiac disorders) | 6 (12)
Pericardial effusion (Cardiac disorders) | 3 (6)
Pericarditis (Cardiac disorders) | 1 (1)
Pulmonary valve disease (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 14 (35)
Supraventricular tachycardia (Cardiac disorders) | 3 (8)
Tricuspid valve disease (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 2 (3)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (5)
Blurred vision (Eye disorders) | 11 (16)
Conjunctivitis (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 7 (10)
Extraocular muscle paresis (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 3 (3)
Eye pain (Eye disorders) | 2 (2)
Eyelid function disorder (Eye disorders) | 1 (1)
Floaters (Eye disorders) | 2 (2)
Photophobia (Eye disorders) | 2 (5)
Watering eyes (Eye disorders) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 6 (9)
Abdominal pain (Gastrointestinal disorders) | 26 (54)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 3 (3)
Anal pain (Gastrointestinal disorders) | 2 (4)
Ascites (Gastrointestinal disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 5 (9)
Colitis (Gastrointestinal disorders) | 6 (9)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 37 (71)
Diarrhea (Gastrointestinal disorders) | 47 (182)
Dry mouth (Gastrointestinal disorders) | 8 (16)
Dyspepsia (Gastrointestinal disorders) | 13 (16)
Dysphagia (Gastrointestinal disorders) | 8 (11)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 4 (6)
Flatulence (Gastrointestinal disorders) | 3 (5)
Gastric hemorrhage (Gastrointestinal disorders) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 13 (22)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 12 (19)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 3 (3)
Hemorrhoids (Gastrointestinal disorders) | 3 (3)
Ileus (Gastrointestinal disorders) | 1 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (8)
Mucositis oral (Gastrointestinal disorders) | 30 (39)
Nausea (Gastrointestinal disorders) | 47 (199)
Oral pain (Gastrointestinal disorders) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (3)
Rectal pain (Gastrointestinal disorders) | 3 (3)
Small intestinal mucositis (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 5 (6)
Toothache (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 40 (106)
Chills (General disorders) | 20 (31)
Edema face (General disorders) | 2 (2)
Edema limbs (General disorders) | 31 (98)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 59 (318)
Fever (General disorders) | 28 (62)
Gait disturbance (General disorders) | 3 (6)
General disorders and administration site conditions - Other, specify (General disorders) | 7 (10)
Infusion related reaction (General disorders) | 4 (4)
Injection site reaction (General disorders) | 1 (1)
Localized edema (General disorders) | 4 (5)
Malaise (General disorders) | 6 (17)
Multi-organ failure (General disorders) | 2 (2)
Neck edema (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 11 (14)
Pain (General disorders) | 16 (42)
Allergic reaction (Immune system disorders) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bronchial infection (Infections and infestations) | 3 (3)
Catheter related infection (Infections and infestations) | 7 (10)
Enterocolitis infectious (Infections and infestations) | 6 (14)
Hepatic infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 18 (31)
Infective myositis (Infections and infestations) | 1 (1)
Joint infection (Infections and infestations) | 1 (5)
Lip infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 14 (33)
Mucosal infection (Infections and infestations) | 6 (9)
Otitis media (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (2)
Phlebitis infective (Infections and infestations) | 1 (1)
Prostate infection (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 3 (3)
Salivary gland infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 5 (7)
Sinusitis (Infections and infestations) | 11 (15)
Skin infection (Infections and infestations) | 7 (18)
Soft tissue infection (Infections and infestations) | 2 (2)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 18 (28)
Urinary tract infection (Infections and infestations) | 14 (30)
Vaginal infection (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 1 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 13 (24)
Fall (Injury, poisoning and procedural complications) | 8 (11)
Fracture (Injury, poisoning and procedural complications) | 2 (2)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 12 (16)
Alanine aminotransferase increased (Investigations) | 48 (204)
Alkaline phosphatase increased (Investigations) | 37 (149)
Aspartate aminotransferase increased (Investigations) | 45 (216)
Blood bilirubin increased (Investigations) | 23 (37)
Cardiac troponin I increased (Investigations) | 5 (6)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 28 (116)
Electrocardiogram QT corrected interval prolonged (Investigations) | 8 (17)
Fibrinogen decreased (Investigations) | 10 (10)
Haptoglobin decreased (Investigations) | 2 (2)
INR increased (Investigations) | 16 (22)
Investigations - Other, specify (Investigations) | 8 (32)
Lymphocyte count decreased (Investigations) | 41 (212)
Lymphocyte count increased (Investigations) | 4 (4)
Neutrophil count decreased (Investigations) | 61 (342)
Platelet count decreased (Investigations) | 63 (413)
Serum amylase increased (Investigations) | 1 (1)
Weight gain (Investigations) | 5 (5)
Weight loss (Investigations) | 11 (121)
White blood cell decreased (Investigations) | 54 (284)
Acidosis (Metabolism and nutrition disorders) | 4 (4)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 33 (98)
Dehydration (Metabolism and nutrition disorders) | 10 (13)
Hypercalcemia (Metabolism and nutrition disorders) | 6 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 51 (284)
Hyperkalemia (Metabolism and nutrition disorders) | 17 (37)
Hypermagnesemia (Metabolism and nutrition disorders) | 21 (32)
Hypernatremia (Metabolism and nutrition disorders) | 15 (25)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 7 (16)
Hyperuricemia (Metabolism and nutrition disorders) | 11 (53)
Hypoalbuminemia (Metabolism and nutrition disorders) | 44 (189)
Hypocalcemia (Metabolism and nutrition disorders) | 45 (129)
Hypoglycemia (Metabolism and nutrition disorders) | 11 (27)
Hypokalemia (Metabolism and nutrition disorders) | 46 (151)
Hypomagnesemia (Metabolism and nutrition disorders) | 28 (80)
Hyponatremia (Metabolism and nutrition disorders) | 38 (122)
Hypophosphatemia (Metabolism and nutrition disorders) | 29 (61)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 3 (29)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (34)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 28 (51)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 14 (35)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 (6)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (15)
Neck pain (Musculoskeletal and connective tissue disorders) | 9 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (38)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 22 (43)
Dysgeusia (Nervous system disorders) | 8 (14)
Dysphasia (Nervous system disorders) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 32 (86)
Hypersomnia (Nervous system disorders) | 1 (2)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 5 (6)
Memory impairment (Nervous system disorders) | 1 (1)
Movements involuntary (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 4 (7)
Neuralgia (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 7 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 25 (118)
Phantom pain (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 3 (5)
Syncope (Nervous system disorders) | 3 (3)
Tremor (Nervous system disorders) | 7 (7)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 20 (56)
Confusion (Psychiatric disorders) | 6 (9)
Delirium (Psychiatric disorders) | 1 (2)
Delusions (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 11 (34)
Hallucinations (Psychiatric disorders) | 4 (6)
Insomnia (Psychiatric disorders) | 28 (51)
Libido decreased (Psychiatric disorders) | 1 (1)
Libido increased (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 2 (2)
Restlessness (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 13 (39)
Bladder spasm (Renal and urinary disorders) | 1 (3)
Chronic kidney disease (Renal and urinary disorders) | 8 (36)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 6 (10)
Proteinuria (Renal and urinary disorders) | 13 (19)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 8 (10)
Urinary frequency (Renal and urinary disorders) | 9 (11)
Urinary incontinence (Renal and urinary disorders) | 3 (6)
Urinary retention (Renal and urinary disorders) | 3 (4)
Urinary tract pain (Renal and urinary disorders) | 3 (7)
Urinary urgency (Renal and urinary disorders) | 3 (3)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Uterine pain (Reproductive system and breast disorders) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 3 (6)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 (13)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (72)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 35 (118)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 (20)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 26 (60)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 (12)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 18 (23)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (12)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 14 (36)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 2 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (30)
Purpura (Skin and subcutaneous tissue disorders) | 6 (12)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (12)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 34 (79)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 16 (56)
Skin induration (Skin and subcutaneous tissue disorders) | 2 (6)
Skin ulceration (Skin and subcutaneous tissue disorders) | 3 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 7 (11)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)
Flushing (Vascular disorders) | 5 (6)
Hematoma (Vascular disorders) | 6 (8)
Hot flashes (Vascular disorders) | 7 (15)
Hypertension (Vascular disorders) | 21 (68)
Hypotension (Vascular disorders) | 16 (27)
Superficial thrombophlebitis (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 7 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT01256398/Prot_SAP_000.pdf